CLINICAL TRIAL: NCT07027553
Title: A Research Study to Understand Whether Remote Exercise Can Improve Physical Activity Levels and Markers of Heart Health in Cystic Fibrosis
Brief Title: Remote Exercise to Improve Physical Activity Levels and Markers of Heart Health in Cystic Fibrosis (RHH-CF)
Acronym: RHH-CF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Rachel McDowell, GW4-CAT PhD Programme for Health Professionals PhD Programme Fellow, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7241-11903
Record Dates: First submitted 2025-05-29; First posted 2025-06-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cystic Fibrosis (CF); Cardiovascular Disease Risk Factors
Keywords: Exercise; Physical activity; Cystic Fibrosis; Cardiovascular disease risk; Mobile health interventions
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Mobile health exercise programme
- Control (Active Comparator)
  Interventions: Other: Lifestyle maintenance

INTERVENTIONS:
Behavioral: Mobile health exercise programme — 8 week personalised exercise intervention. Delivered and monitored via mobile health technology
  Arms: Intervention
Other: Lifestyle maintenance — Continue current lifestyle
  Arms: Control

SUMMARY:
With advances in genetic therapies, many people with Cystic Fibrosis (CF) are living longer. With the improvement in life expectancy has emerged an increased risk of cardiovascular disease (CVD). Factors such as insulin resistance, reduced physical activity, rising blood pressure from newer medications, and changes in body mass index have made cardiovascular health a growing concern in CF care.

This study aims to assess whether a remotely delivered, monitored exercise programme can increase physical activity levels in adults with CF. Secondary outcomes will explore whether the intervention improves key CVD risk factors. Participants will be randomly assigned to either a control group or an intervention group, which will complete an 8-week home-based aerobic and resistance exercise programme. Exercise intensity will be tailored using the Rate of Perceived Exertion scale.

Key outcomes include weekly physical activity levels, body mass index, waist circumference, lung function (spirometry) and blood biomarkers. Home-based capillary blood tests, analysed pre- and post-intervention, will measure cholesterol, lipid profiles, inflammation and other relevant hormones.

ELIGIBILITY:
Inclusion Criteria:

* Past diagnosis of Cystic Fibrosis confirmed via two copies of a faulty CFTR gene, or; previous sweat chloride test with a result >60mmol/L chloride, or; prescribed modulator therapy (Orkambi, Symkevi, Kaftrio);

Exclusion Criteria:

* Any reported condition, behaviour or reported use of substances which may pose undue personal risk to the participant or introduce bias into the study, except for any which are ubiquitous in society and so would be equally distributed between groups and/or therefore relevant to generalisation (e.g. caffeine)
* Medications which increase risk of harm to a participant exercising remotely such as fluoroquinolone antibiotics, beta blockers, or blood pressure medication
* Individuals with unstable or poorly controlled diabetes
* Individuals on statins
* Females who are pregnant or lactating
* Individuals with a previous self-reported history of an eating disorder
* Individuals unable to provide informed consent e.g. inability to read or speak English
* Individuals who are not weight stable (i.e. >3kg change in body mass in the past 3 months)
* Individuals awaiting a solid organ transplant, have a diagnosis of pulmonary hypertension or require long term oxygen therapy to exercise at home
* Individuals with chest pain, dizziness or loss of consciousness during exercise, who have been instructed by a doctor to only do certain types/quantity of physical activity
* Individuals on any current ongoing medication or treatment for injuries or illness which impact on their ability to do physical tasks or exercises
* Individuals who are PAR-Q positive response during screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-19 (Estimated); Primary Completion 2026-05-19 (Estimated); Study Completion 2026-09-19 (Estimated)

PRIMARY OUTCOMES:
Weekly minutes of moderate-vigorous physical activity | Baseline and 8 weeks
  Measured using a Geneactiv wrist-based activity monitor

SECONDARY OUTCOMES:
Body mass index | Baseline and 8 weeks
  kg/m2
Waist circumference | Baseline and 8 weeks
  Measured in centimetres
Waist to hip ratio | Baseline and 8 weeks
  Measured in centimetres
1-minute sit to stand test | Baseline and 8 weeks
  Participant stands up and sits down from a chair for one minute and the number of completed sit-to-stands is recorded.
Multidimensional Fatigue Inventory | Baseline and 8 weeks
  Measured on 20 questions with a scale of 1-5. The maximum possible score is 100 with a higher score indicating more acute levels of fatigue
Cystic Fibrosis Questionnaire Revised | Baseline and 8 weeks
  Quality of life questionnaire validated for Cystic Fibrosis. Scores range from 0 to 100, with higher scores indicating better health.
Manchester Musculoskeletal Screening tool | Baseline and 8 weeks
  Musculoskeletal pain questionnaire. A higher score indicates a worse outcome. Maximum possible score is 50, minimum possible score is 0
Sleep quality | Baseline and 8 weeks
  3-day sleep quality and quantity diary
Fasting insulin levels, pmol/L | Baseline and 8 weeks
  Taken from the early morning fasted capillary blood sample
Fasting triglyceride concentration, mmol/L | Baseline and 8 weeks
  Taken with the early morning fasted capillary blood sample
Serum fructosamine, mmol/L | Baseline and 8 weeks
  Taken from the fasted early morning capillary blood sample
Fasting LDL-C, HDL-C and total cholesterol, mmol/L | Baseline and 8 weeks
  Taken from the fasted early morning capillary blood samples
High sensitivity C-reactive protein, mg/L | Baseline and 8 weeks
  Measured in the capillary blood samples taken
Forced expiratory volume in one second | Baseline and 8 weeks
  Obtained by spirometry. Recorded as litres per minute and percentage predicted values using Global Lung Index reference values
Forced Vital Capacity | Baseline and 8 weeks
  Obtained through spirometry. Recorded as litres per minute and percentage predicted values using Global Lung Index reference values.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Nutrition, Exercise and Metabolism, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available open access on the University of Bath Research Data Archive (RDA) at the point of publication in a peer-reviewed journal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: These will become available at the point of publication permanently.
URL: https://researchdata.bath.ac.uk/

REFERENCES:
- See also: Related Info — https://www.bath.ac.uk/research-centres/centre-for-nutrition-exercise-and-metabolism/